CLINICAL TRIAL: NCT01523990
Title: A Study in Healthy Volunteers to Evaluate the Safety, Tolerability, and Pharmacokinetics Profiles of Single and Multiple Ascending Oral Doses of TG-2349, and Followed by a Dose-Ranging Study in Hepatitis C Genotype 1 Infected Patients
Brief Title: A Study to Evaluate the Safety, Tolerability, and PK in Healthy Volunteers and HCV Genotype 1 Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TaiGen Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TG-2349-01
Record Dates: First submitted 2011-10-13; First posted 2012-02-01 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Healthy; Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (27):
- Panel I (TG-2349) (Experimental): Sequential single oral dose taken by healthy East and Caucasian volunteers from 50 mg (fasted) to 50 mg (fed) of TG-2349 with 1 week follow-up after each dosage. A washout period of at least 10 days between the 1st and the 2nd dose is required.
  Interventions: Drug: TG-2349
- Panel I (placebo) (Placebo Comparator): Sequential single oral dose taken by healthy East and Caucasian volunteers from 50 mg (fasted) to 50 mg (fed) of placebo with 1 week follow-up after each dosage. A washout period of at least 10 days between the 1st and the 2nd dose is required.
  Interventions: Drug: placebo
- Panel II (TG-2349) (Experimental): Sequential single oral dose taken by healthy East and Caucasian volunteers from 100 mg (fasted) to 100 mg (fed) of TG-2349 with 1 week follow-up after each dosage. A washout period of at least 10 days between the 1st and the 2nd dose is required.
  Interventions: Drug: TG-2349
- Panel II (placebo) (Placebo Comparator): Sequential single oral dose taken by healthy East and Caucasian volunteers from 100 mg (fasted) to 100 mg (fed) of placebo with 1 week follow-up after each dosage. A washout period of at least 10 days between the 1st and the 2nd dose is required.
  Interventions: Drug: placebo
- Panel III (TG-2349) (Experimental): Sequential single oral dose taken by healthy East and Caucasian volunteers from 200 mg (fasted or fed) to 400 mg (fasted or fed) of TG-2349 with 1 week follow-up after each dosage. A washout period of at least 10 days between the 1st and the 2nd dose is required.
  Interventions: Drug: TG-2349
- Panel III (placebo) (Placebo Comparator): Sequential single oral dose taken by healthy East and Caucasian volunteers from 200 mg (fasted or fed) to 400 mg (fasted or fed) of placebo with 1 week follow-up after each dosage. A washout period of at least 10 days between the 1st and the 2nd dose is required.
  Interventions: Drug: placebo
- Panel IV (TG-2349) (Experimental): Sequential single oral dose taken by healthy East and Caucasian volunteers from 600 mg (fasted or fed) to 800 mg (fasted or fed) of TG-2349 with 1 week follow-up after each dosage. A washout period of at least 10 days between the 1st and the 2nd dose is required.
  Interventions: Drug: TG-2349
- Panel IV (placebo) (Placebo Comparator): Sequential single oral dose taken by healthy East and Caucasian volunteers from 600 mg (fasted or fed) to 800 mg (fasted or fed) of placebo with 1 week follow-up after each dosage. A washout period of at least 10 days between the 1st and the 2nd dose is required.
  Interventions: Drug: placebo
- Panel V (TG-2349) (Experimental): Oral dose taken once daily for 5 consecutive days at dose level of 100 mg taken by healthy East and Caucasian volunteers .
  Interventions: Drug: TG-2349
- Panel V (placebo) (Placebo Comparator): Oral dose taken once daily for 5 consecutive days at dose level of 100 mg taken by healthy East and Caucasian volunteers .
  Interventions: Drug: placebo
- Panel VI (TG-2349) (Experimental): Oral dose taken once daily for 5 consecutive days at dose level of 200 mg taken by healthy East and Caucasian volunteers .
  Interventions: Drug: TG-2349
- Panel VI (placebo) (Placebo Comparator): Oral dose taken once daily for 5 consecutive days at dose level of 200 mg taken by healthy East and Caucasian volunteers .
  Interventions: Drug: placebo
- Panel VII (TG-2349) (Experimental): Oral dose taken once daily for 5 consecutive days at dose level of 400 mg taken by healthy East and Caucasian volunteers .
  Interventions: Drug: TG-2349
- Panel VII (placebo) (Placebo Comparator): Oral dose taken once daily for 5 consecutive days at dose level of 400 mg taken by healthy East and Caucasian volunteers .
  Interventions: Drug: placebo
- Panel VIII (TG-2349) (Experimental): Oral dose taken once daily for 5 consecutive days at dose level of 600 mg taken by healthy East and Caucasian volunteers .
  Interventions: Drug: TG-2349
- Panel VIII (placebo) (Placebo Comparator): Oral dose taken once daily for 5 consecutive days at dose level of 600 mg taken by healthy East and Caucasian volunteers .
  Interventions: Drug: placebo
- Panel IX (TG-2349) (Experimental): Oral dose taken once daily for 3 consecutive days at dose level of 200 mg (fed) taken by HCV genotype 1 (including subtypes 1a or 1b or mixed 1a/1b) infected patients.
  Interventions: Drug: TG-2349
- Panel IX (placebo) (Placebo Comparator): Oral dose taken once daily for 3 consecutive days at dose level of 200 mg (fed) taken by HCV genotype 1 (including subtypes 1a or 1b or mixed 1a/1b) infected patients.
  Interventions: Drug: placebo
- Panel X (TG-2349) (Experimental): Oral dose taken once daily for 3 consecutive days at dose level of 400 mg (fed) taken by HCV genotype 1 (including subtypes 1a or 1b or mixed 1a/1b) infected patients.
  Interventions: Drug: TG-2349
- Panel X (placebo) (Placebo Comparator): Oral dose taken once daily for 3 consecutive days at dose level of 400 mg (fed) taken by HCV genotype 1 (including subtypes 1a or 1b or mixed 1a/1b) infected patients.
  Interventions: Drug: placebo
- Panel XI (TG-2349) (Experimental): Oral dose taken once daily for 3 consecutive days at dose level of 600 mg (fed) taken by HCV genotype 1 (including subtypes 1a or 1b or mixed 1a/1b) infected patients.
  Interventions: Drug: TG-2349
- Panel XI (placebo) (Placebo Comparator): Oral dose taken once daily for 3 consecutive days at dose level of 600 mg (fed) taken by HCV genotype 1 (including subtypes 1a or 1b or mixed 1a/1b) infected patients.
  Interventions: Drug: placebo
- Panel XII (TG-2349) (Experimental): Oral dose taken once daily for 3 consecutive days at dose level of 600 mg (fed) taken by HCV genotype 2 infected, treatment-naive patients.
  Interventions: Drug: TG-2349
- Panel XIII (TG-2349) (Experimental): Oral dose taken once daily for 3 consecutive days at dose level of 600 mg (fed) taken by HCV genotype 3 infected, treatment-naive patients.
  Interventions: Drug: TG-2349
- Panel XIV (TG-2349) (Experimental): Oral dose taken once daily for 3 consecutive days at dose level of 600 mg (fed) taken by HCV genotype 4 infected, treatment-naive patients.
  Interventions: Drug: TG-2349
- Panel XV (TG-2349) (Experimental): Oral dose taken once daily for 3 consecutive days at dose level of 600 mg (fed) taken by HCV genotype 5 infected, treatment-naive patients.
  Interventions: Drug: TG-2349
- Panel XVI (TG-2349) (Experimental): Oral dose taken once daily for 3 consecutive days at dose level of 600 mg (fed) taken by HCV genotype 6 infected, treatment-naive patients.
  Interventions: Drug: TG-2349

INTERVENTIONS:
Drug: TG-2349 — Supplied as oral liquid formulation in pre-filled glass syringe. Two dose strengths, 25 mg TG-2349 (25 mg/mL in PEG 400, 1.1 mL fill) and 200 mg TG-2349 (50 mg/mL in PEG 400, 4.1 mL fill), are filled into 5-mL type 1 glass syringes. Required doses during clinical study are to be dispensed using the combination of the two dose units. The entire content of the syringe is to be taken by mouth.
  Arms: Panel I (TG-2349); Panel II (TG-2349); Panel III (TG-2349); Panel IV (TG-2349); Panel IX (TG-2349); Panel V (TG-2349); Panel VI (TG-2349); Panel VII (TG-2349); Panel VIII (TG-2349); Panel X (TG-2349); Panel XI (TG-2349); Panel XII (TG-2349); Panel XIII (TG-2349); Panel XIV (TG-2349); Panel XV (TG-2349); Panel XVI (TG-2349)
Drug: placebo — Available in two different unit doses, 1.1 mL and 4.1 mL PEG 400 in 5-mL type 1 glass syringes. They are identical in appearance and similar in weight to TG-2349 oral liquid syringes.
  Arms: Panel I (placebo); Panel II (placebo); Panel III (placebo); Panel IV (placebo); Panel IX (placebo); Panel V (placebo); Panel VI (placebo); Panel VII (placebo); Panel VIII (placebo); Panel X (placebo); Panel XI (placebo)

SUMMARY:
A Safety Study to Evaluate the Safety, Tolerability, and Pharmacokinetics in HCV Genotype 1 Infected Patients

DETAILED DESCRIPTION:
A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study in Healthy East Asian and Caucasian Volunteers to Evaluate the Safety, Tolerability, and Pharmacokinetics Profiles of Single and Multiple Ascending Oral Doses of TG-2349, and Followed by a Dose-Ranging Study in Hepatitis C Genotype 1 Infected Patients.

ELIGIBILITY:
Inclusion Criteria:

* East Asian or Caucasian subjects, male or female, and 18 to 65 years of age inclusive
* Body mass index (BMI) in the range of 19.0 to 30.0 kg/m2 and body weight ≥ 50 kg inclusive
* In generally good physical and mental health status on the basis of a medical history review, medical evaluation including vital signs and physical examination, 12-lead ECG, and laboratory results at screening
* For females, one of the following criteria must be fulfilled:

  1. At least 1 year post menopausal, or
  2. Surgically sterile, or
  3. Willing to use a double barrier method [intrauterine device (IUD) plus condom, spermicidal gel plus condom] of contraception from screening until 30 days after the last dose of study drug
* Males must be willing to use a reliable form of contraception (use of a condom or a partner fulfilling the above criteria) from screening until 30 days after the last dose of study drug
* Willing to abstain from caffeine- or xanthine-containing beverages, including coffee and tea, alcohol, grapefruit juice, and Seville oranges during the stay-on-site period
* Willing and able to provide written informed consent

Exclusion Criteria:

* Positive serological test for IgM anti-HAV antibody, HBsAg or anti-HCV antibody at screening
* Positive ELISA test for HIV-1 or HIV-2 at screening
* Any abnormal laboratory values at screening: Hemoglobin (Hb) <12.0g/dL for women and <13.0g/dL for men, white blood cell count (WBC) <3,000 cells/mm3, absolute neutrophil count <1,500 cells/mm3, platelet count <100,000 cells/mm3, serum creatinine ≥ 2 mg/dL, ALT or AST levels ≥ 2 xULN, total bilirubin

  ≥ 1.5 x ULN, INR (International Normalized Ratios for prothrombin time) ≥ 1.5 xULN
* Any abnormal laboratory values that are considered clinically significant by the Investigator at screening
* QTcF greater than 450 msec for females and 430 msec for males at screening
* History of renal, hepatic impairment, stomach or intestinal surgery or resection, malabsorption syndrome
* History of seizures, epilepsy, cardiovascular, diabetes or cancer (except basal cell carcinoma)
* History or family history of prolonged QT interval or family history of sudden cardiac death at a young age
* History of drug allergy or hypersensitivity, especially to sulfa drugs
* History or evidence of abuse of alcohol, barbiturate, amphetamine, recreational or narcotic drug use within 6 months prior to first dose of study drug administration
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of a psychiatric illness, or have any history of suicide attempt or depression
* Anemia or blood/plasma donation within 30 days prior to first dose of study drug administration
* Pregnant or breast-feeding
* Use of tobacco or nicotine-containing products within 30 days prior to first dose of study drug administration
* Use of concomitant medication, including herbal remedies, and dietary supplements (except for paracetamol/acetaminophen, ibuprofen and hormonal contraceptives) within 14 days prior to first dose of study drug administration
* Received any other investigational drug within 30 days prior to first dose of study drug administration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) profiles of single and multiple ascending oral doses of TG-2349 in healthy East Asian and Caucasian volunteers. | predose, and 1,2,3,4,6,8,12,24,36,48,72,96 hours post-dose
  Dose proportionality will be assessed by evaluating PK parameters AUC0-t, AUC0-inf, and Cmax. Parameters that are not dose dependent will be assessed by evaluating Tmax, t1/2, and λz. The linear relationship between the log-transformed PK parameter and the natural log of the dose will be tested using a linear lack-of-fit test. The dose-dependent parameters will not be dose normalized. Residual analysis will be used to assess the assumptions of normality and variance homogeneity for the statistical model.
Safety and tolerability of single and multiple ascending oral doses of TG-2349 in healthy East Asian and Caucasian volunteers. | predose, and 2,4,6,8,12,24,48,72,96 hours post-dose
  Vital signs, physical examinations, 12-lead ECG, safety laboratory parameter abnormalities, and other toxicities graded by the National Cancer Institute (NCI) Common Toxicity Criteria (CTC) version 4.0 will be examined to evaluate safety profiles of the study treatments. Special attention will be paid to Grade III or IV toxicities in all treatment levels.
Pharmacokinetics (PK) profiles of multiple oral doses of TG-2349 in genotype 1, 2, 3, 4, 5, and 6 HCV-infected patients. | predose, and 1,2,3,4,6,8,12,24,36,48,72,96 hours post-dose
  Dose proportionality will be assessed by evaluating PK parameters AUC0-t, AUC0-inf, and Cmax. Parameters that are not dose dependent will be assessed by evaluating Tmax, t1/2, and λz. The linear relationship between the log-transformed PK parameter and the natural log of the dose will be tested using a linear lack-of-fit test. The dose-dependent parameters will not be dose normalized. Residual analysis will be used to assess the assumptions of normality and variance homogeneity for the statistical model.
Safety and tolerability of multiple ascending oral doses of TG-2349 in genotype 1, 2, 3, 4, 5, and 6 HCV-infected patients. | predose, and 4,6,12 hours post-dose
  Vital signs, physical examinations, 12-lead ECG, safety laboratory parameter abnormalities, and other toxicities graded by the National Cancer Institute (NCI) Common Toxicity Criteria (CTC) version 4.0 will be examined to evaluate safety profiles of the study treatments. Special attention will be paid to Grade III or IV toxicities in all treatment levels.
Antiviral activity of multiple ascending oral doses of TG-2349 in genotype 1, 2, 3, 4, 5, and 6 HCV-infected patients. | predose, and 1,2,3,4,6,8,12,24,36,48,72,96 hours post-dose
  Descriptive statistics and graphs will be presented for the antiviral variables. Change from pre dose will be analyzed descriptively for each time point after study drug administration. Graphic displays of raw data and changes over time will be performed at each dosing level (plots of raw data of TG-2349 at each time point with mean and median).
  The breakthrough is defined as a greater than or equal to 1 log10 increase in HCV RNA above nadir, or detectable HCV RNA, while on treatment, after an initial drop to a level of below the detection. The slope of the plasma viral RNA decrease during the first few days of treatment, any subsequent plasma viral RNA increase observed during and/or after dosing, and all breakthrough events should be recorded and summarized.

SECONDARY OUTCOMES:
The food effect of TG-2349 in healthy volunteers. | 1 week
  Food effect will be evaluated at two lower doses of 50 mg and 100 mg in panel I and panel II of the study.The primary PK parameters to investigate the food effect are AUC0-inf, AUC0-24, and Cmax. The secondary PK parameters to investigate the food effect are Tmax, t½, CL.
Appearance of viral variants if any in genotype 1, 2, 3, 4, 5, and 6 HCV-infected patients. | during and after 3 days of TG-2349 dosing, the 4-week and 1 year follow-up periods
  Appearance of phenotype and genotype variants potentially arising during the 3-day treatment period and during the 4-week and 1 year follow-up periods.
Ethnicity differences in safety and tolerability between East Asian and Caucasian volunteers. | predose, and 2,4,6,8,12,24,48,72,96 hours post-dose
  Vital signs, physical examinations, 12-lead ECG, safety laboratory parameter abnormalities, and other toxicities graded by the National Cancer Institute (NCI) Common Toxicity Criteria (CTC) version 4.0 will be examined to evaluate safety profiles of the study treatments. Special attention will be paid to Grade III or IV toxicities in all treatment levels.
Ethnicity differences in Pharmacokinetics (PK) profiles between East Asian and Caucasian volunteers. | predose, and 1,2,3,4,6,8,12,24,36,48,72,96 hours post-dose
  Dose proportionality will be assessed by evaluating PK parameters AUC0-t, AUC0-inf, and Cmax. Parameters that are not dose dependent will be assessed by evaluating Tmax, t1/2, and λz. The linear relationship between the log-transformed PK parameter and the natural log of the dose will be tested using a linear lack-of-fit test. The dose-dependent parameters will not be dose normalized. Residual analysis will be used to assess the assumptions of normality and variance homogeneity for the statistical model.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Sims, DO, Principal Investigator — WCCT
Locations (1):
- WCCT, Cypress, California, United States